CLINICAL TRIAL: NCT02286778
Title: The Eradication of Malignant Carcinoma in the Breast Tissue Using an ATP (Adenosine-5'-Triphosphate) Inhibitor
Brief Title: Eradication of Malignant Carcinoma in the Breast Tissue
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Optimal Health Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: F-9892131B
Record Dates: First submitted 2014-11-03; First posted 2014-11-10 (Estimated); Last update posted 2017-08-03 (Actual); Status verified 2017-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Acetogenins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Acetogenins (Active Comparator): Dietary Supplement: Acetogenins BID for 12 months
  Interventions: Dietary Supplement: Acetogenins
- Placebo (Placebo Comparator): Dietary Supplement: No Acetogenins BID for 12 months
  Interventions: Dietary Supplement: Placebo
- Control (No Intervention): Control subjects will not receive the Acetogenins or the placebo. They will be evaluated every other month to monitor disease progress.

INTERVENTIONS:
Dietary Supplement: Acetogenins — Acetogenins BID for 12 months
  Arms: Acetogenins
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to confirm the findings of an early study and expand our knowledge of treating Malignant Carcinoma in the Breast Tissue Using an ATP (Adenosine-5'-Triphosphate) Inhibitor.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of breast cancer
* Referred to the study by their treating physician

Exclusion Criteria:

* Any type of treatment for breast cancer before starting the study

Ages: 35 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-02; Primary Completion 2017-01 (Actual); Study Completion 2017-08-01 (Actual)

PRIMARY OUTCOMES:
Number of participants tumor free | 12 months
  assessed by MRI

CONTACTS AND LOCATIONS:
Overall Officials: John A Shaw, MD, Principal Investigator — Optimal Health Research; Steven Osguthorpe, ND, Principal Investigator — Optimal Health Research